CLINICAL TRIAL: NCT04504240
Title: Role of Famotidine in the Clinical Recovery and Symptomatic Improvement of COVID-19 Patients.
Brief Title: Role of Famotidine in the Clinical Improvement of COVID-19 Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chattogram General Hospital (Other Government)
Collaborators: M Abdur Rahim Medical College and Hospital (Other Government); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Abu Taiub Mohammed Mohiuddin Chowdhury, Doctoral Resident, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000753/980
Record Dates: First submitted 2020-08-06; First posted 2020-08-07 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Covid19
Keywords: COVID 19; Famotidine; Bangladesh
MeSH Terms: conditions — COVID-19 | interventions — Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: FAMOTIDINE treatment group (Experimental): FAMOTIDINE 40mg to 60mg 8hourly in an empty stomach along with other treatments.
  Interventions: Drug: Famotidine 20 MG
- Group B: Control group (Active Comparator): Treatment as given with a PPI.
  Interventions: Drug: Famotidine 20 MG

INTERVENTIONS:
Drug: Famotidine 20 MG — Famotidine; tablet Famotac 20mg oral form.
  Other Names: Famotac 20mg

SUMMARY:
This study is aimed to investigate the effect of Famotidine in the clinical recovery of COVID-19 patients. COVID19 is a worldwide pandemic. Hence SARS-CoV-2 is a novel virus; there is no specific medication against it. Like other countries of the world, Besides antiviral drugs, immunosuppressive agents, and symptomatic therapy like H2 receptor blocker FAMOTIDINE came to the limelight due to its role in reducing the symptoms of COVID-19 patients. The study will include COVID-19 participants to confirm by RT PCR or an HRCT chest. Detail history of each participant with comorbidity will be taken and will be examined carefully. The hospitalized patients admitted to the HDU/ICU units will be enrolled in this study. Critically ill patients who require ventilator support will not be included in this study. The outcome of the Famotidine treatment will be evaluated and compared with a control group.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection confirmed by RT PCR or CT Chest.
* Severe COVID-19 patients require hospitalization under HDU/ICU.

Exclusion Criteria:

* Patients with severe and/or uncontrolled medical conditions with significantly compromised organ function.
* Patients who were hospitalized from the before due to other reasons.
* Contraindication / possible drug interaction with Famotidine with existing therapy.
* Immunocompromised patients.
* Pregnancy, Pulmonary Tuberculosis, AIDS

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Time to Clinical Improvement (TTCI) | Following randomization 30days.
  Time to clinical improvement (TTCI) was defined as time from randomization to National Early Warning Score 2 (NEWS2) Score of ≤2 maintained for 24 Hours.
Time to symptomatic recovery. | Following randomization 30 days.
  Time to Symptomatic recovery was defined as the duration (in days) that required for the relief of the COVID-19 symptoms from the day of hospitalization.

SECONDARY OUTCOMES:
Mortality Rate | Following randomization 30 days.
  Mortality Rate in percentage in study groups.
Duration of ICU Stay. | Following randomization 30 days.
  Duration of ICU Stay in days.
Total hospital stay. | Following randomization 30 days.
  Time from randomization to hospital discharge or "Ready for discharge" (as evidenced by normal body temperature and respiratory rate, and stable oxygen saturation on ambient Air or ≤4L supplemental oxygen).
Time to clinical failure or death. | Following randomization 30 days.
  Time to clinical failure, defined as the time from randomization to the first occurrence of death, mechanical ventilation or withdrawal (whichever occurs first).
Time to Viral clearance / COVID-19 recovery. | Following randomization 60 days.
  This was defined as the duration (in days) from the first positive PCR to the first negative PCR (Confirmed by a repeat negative PCR after 7days) for SARS-Cov-2 infection following hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Abu Taiub Mohammed Mohiuddin Chowdhury, MBBS, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (2):
- Bangladesh (2):
  - Chattogram General Hospital, Chittagong
  - M. Abdur Rahim Medical College Hospital, Dinājpur

IPD SHARING:
Plan to Share IPD: No